CLINICAL TRIAL: NCT04458558
Title: Improving Access to Abortion in the Republic of Georgia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Information and Counseling on Reproductive Health - Tanadgoma (Other)
Collaborators: Gynuity Health Projects (Other); Healthy Life (Unknown); Grand Challenges Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2.1
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Abortion Early; Pregnancy Related
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Intervention Model Description: Prospective Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical abortion patients (Experimental): Oral mifepristone 200 mg followed by misoprostol 800 mcg administered buccally (at 24-48 hours following mifepristone).
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — Participants will receive mifepristone at a preferred address by mail rather than standard care at clinic visit.

SUMMARY:
In the Republic of Georgia, the medical abortion regimen involves three in-person visits. This study aims to pilot and evaluate a simplified medical abortion service delivery model that will reduce the number of in-person visits to only one visit for diagnosis and counseling. Medication will be mailed along with two multi-level pregnancy tests to study participants, who will assess their abortion outcome at home.

DETAILED DESCRIPTION:
This prospective cohort study of patients obtaining medical abortion medications by mail. The study investigators aim to recruit approximately 120 patients for this study across three study sites that have extensive experience providing early medical abortion. Five days after undergoing in-person consultation and necessary exams to assess eligibility for medical abortion, study team will mail study participants medical abortion pills and two multi-level urine pregnancy tests. Medical abortion follow-up will occur at the participant's home approximately two weeks after the initial visit, and the multi-level pregnancy test will be used to assess abortion outcome. At follow-up, study participants will be asked questions about the results of the multi-level pregnancy test, and their experience and feedback about the acceptability of the process. At the conclusion of the study, investigators will interview providers to better undertand their experience with the simplified medical abortion service delivery model.

ELIGIBILITY:
Inclusion Criteria:

* Women seeking medical abortion through 58 days gestation
* Eligible for medical abortion according to study provider's assessment
* Able to receive physical mail
* Have access to a phone
* Be willing and able to consent to participate in the study
* Be willing to follow study procedures

Exclusion Criteria:

* Not seeking medical abortion
* Contraindications to medical abortion

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who report satisfactory experience | Day 14 following initial medical abortion visit
  Number of participants who report being "satisfied" or "very satisfied" with the simplified medical abortion service delivery model
Number of providers who report satisfactory experience | End of the study, month 15
  Number of providers who report being "satisfied" or "very satisfied" with the simplified medical abortion service delivery model

SECONDARY OUTCOMES:
Number of participants with adverse event | Up to 6 weeks after initial medical abortion visit
  Number of participants who had a medical problem that required them to go to the hospital, emergency department or a doctor's office (other than regularly scheduled follow-up visit) since receiving medical abortion pills
Number of participants with a complete abortion with medication alone and who do not require additional interventions to complete the procedure | Up to 6 weeks after initial medical abortion visit
  Number of participants who report that their abortion is complete as assessed by the multi-level pregnancy test and medical history.
Number of particpants with adverse event associated with mailing of medical abortion medications | Up to 6 weeks after initial medical abortion visit
  Number of participants who had a problem (such as delayed and lost packages) receiving medical abortion medications by mail
Cost associated with the simplified medical abortion service delivery model | Up to 6 weeks after initial medical abortion visit
  Cost savings associated with participant travel to the clinic and cost of the standard care at the clinic.
Number of participants who refuse to receive medical abortion pills by mail | End of the study, month 15
  Number of participants who refuse to receive medical abortion pills by mail during the study period

CONTACTS AND LOCATIONS:
Locations (3):
- Georgia (3):
  - Batumi Medical Center, Batumi
  - David Gagua Clinic, Tbilisi
  - Clinic Elite, Zestaponi

IPD SHARING:
Plan to Share IPD: No